CLINICAL TRIAL: NCT02359292
Title: Cross-over Clinical Pharmacology Study, to Evaluate the Total Systemic Exposure and Lung Bioavailability of CHF 5993 pMDI Combination Across Two Different Dose Strengths, Administered With and Without Activated Charcoal, in Healthy Volunteers
Brief Title: Clinical Pharmacology Study to Evaluate the Total Systemic Exposure and Lung Bioavailability of CHF 5993 pMDI Combination in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-05993AB2-01
Record Dates: First submitted 2015-01-30; First posted 2015-02-10 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- CHF 5993 HS 200/6/25 pMDI (Experimental): High Strength fixed combination
  Interventions: Drug: CHF 5993 HS 200/6/25 pMDI
- CHF 5993 MS 100/6/25 pMDI (Active Comparator): Medium Strength fixed combination
  Interventions: Drug: CHF 5993 MS 100/6/25 pMDI
- CHF 5993 HS 200/6/25 pMDI + Charcoal Block (Experimental): High Strength fixed combination plus Charcoal Block
  Interventions: Drug: CHF 5993 HS 200/6/25 pMDI + Charcoal Block
- CHF 5993 MS 100/6/25 pMDI + Charcoal Block (Active Comparator): Medium Strength fixed combination plus Charcoal Block
  Interventions: Drug: CHF 5993 MS 100/6/25 pMDI + Charcoal Block
- Placebo pMDI (Placebo Comparator): Placebo
  Interventions: Drug: Placebo pMDI

INTERVENTIONS:
Drug: CHF 5993 HS 200/6/25 pMDI
  Arms: CHF 5993 HS 200/6/25 pMDI
Drug: CHF 5993 MS 100/6/25 pMDI
  Arms: CHF 5993 MS 100/6/25 pMDI
Drug: CHF 5993 HS 200/6/25 pMDI + Charcoal Block
  Arms: CHF 5993 HS 200/6/25 pMDI + Charcoal Block
Drug: CHF 5993 MS 100/6/25 pMDI + Charcoal Block
  Arms: CHF 5993 MS 100/6/25 pMDI + Charcoal Block
Drug: Placebo pMDI
  Arms: Placebo pMDI

SUMMARY:
The study is performed to evaluate the total systemic exposure and lung bioavailability of CHF 5993 pMDI combination, in healthy volunteers subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study related procedure.
2. Able to understand the study procedures, the risks involved and ability to be trained to use the devices correctly.
3. Male and female subjects aged 18 to 55 years inclusive.
4. Body mass index (BMI) within the range of 18 to 30 kg/m2 inclusive.
5. Non- or ex-smokers who smoked < 5 pack years (pack-years = the number of cigarette packs per day, times the number of years) and stopped smoking > 1 year prior to screening.
6. Good physical and mental status, determined on the basis of the medical history and a general clinical examination, at screening and before randomization.
7. Lung function measurements within normal limits (Normal values (according to GINA 2014 document): FEV1/FVC > 0.70 and FEV1 > 80% predicted).
8. Male subjects: they and/or their partner must be willing to use an approved method of contraception from the time of screening and until 30 days after the last dose of study. Subjects must not donate sperm for 30 days after the last dose of study drug.*
9. Female subjects: post-menopausal women having at least 12 months of natural (spontaneous) amenorrhea, or women of childbearing potential (defined as all women physiologically capable of becoming pregnant), using an acceptable method of contraception
10. Surgical sterilization (i.e. bilateral tubal ligation, hysterectomy for females; vasectomy for males)
11. Hormonal contraception (implantable, injectable, patch, oral)
12. Double-barrier methods: condom and occlusive cap (diaphragm or cervical/vault caps)
13. Placement of an intrauterine device (IUD) or intrauterine system (IUS).

Exclusion Criteria:

1. Blood donation (equal or more than 450 ml) or blood loss, less than 8 weeks before inhalation of the study medication.
2. Female subjects: pregnant or lactating women (where pregnancy is defined as the state of a female after conception and until the termination of the gestation) confirmed by a positive urine test at screening and randomization.
3. Positive HIV1 or HIV2 serology.
4. Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C.
5. Unsuitable veins for repeated venipuncture.
6. History of alcohol abuse within 12 months prior to screening.
7. History of drug abuse within 12 months prior to screening (or positive urine drug test performed at screening).
8. Subjects who have a positive urine test for cotinine.
9. Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical investigation. Note: In case of abnormal laboratory values, the test can be performed again once before randomization.
10. Clinically relevant and uncontrolled hepatic, gastrointestinal, endocrine, metabolic, neurologic, or psychiatric disorder that may interfere with successful completion of this protocol.
11. History of glaucoma, symptomatic prostatism or urinary retention.
12. Subjects who have cardiovascular condition such as, but not limited to, unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, acute ischemic heart disease in the last year prior to study screening, history of sustained cardiac arrhythmias or sustained and non-sustained cardiac arrhythmias diagnosed in the last 6 months (sustained means lasting more than 30 seconds and or ending only with external action, and or leads to hemodynamic collapse; non-sustained means > 3 beats < 30 seconds, and or ending spontaneously, and or asymptomatic), impulse conduction high degree blocks, ICD implant
13. Abnormal ECG (i.e.: QRS > 120 msec, PR > 220 msec, HR < 40 bpm, HR > 110 bpm, QTcF > 450 ms for males or QTcF > 470 ms for females) at screening.

    Note: In case of abnormal ECG, the test can be performed again once before randomization.
14. Clinically significant abnormal 24h-Holter monitoring at screening (if necessary the Holter evaluation can be done on another day before randomization).
15. Abnormal Blood Pressure (Average Diastolic Blood Pressure > 90 mmHg or average Systolic Blood Pressure > 140 mmHg) at screening.

    Note: In case of abnormal blood pressure, measure can be done again once before randomization.
16. Participation in another clinical trial where investigation drug was received less than 8 weeks prior to screening.
17. History of hypersensitivity to any of the excipients contained in the formulations used in the trial.
18. Subject taking any drug treatment, including prescribed or OTC medicines as well as vitamins, homeopathic remedies etc, taken in the 14 days before the screening with the exception of :

    1. Occasional paracetamol (maximum 2 g per day with a maximum of 10 g per 14 days for mild non-excluding conditions);
    2. Hormonal contraceptives;
    3. Hormonal replacement treatment for post-menopausal women.
19. Subject taking treatment, with enzyme-inducing or enzyme-inhibiting drugs and biologic drugs and with any drug known to have a well-defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole), taken since 3 months before screening until randomization.
20. Heavy caffeine drinker (> 5 caffeinated beverages e.g., coffee, tea, cola per day).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Systemic exposure of B17MP, Formoterol and Glycopyrronium bromide, without charcoal block (To evaluate the total systemic exposure as AUCt and Cmax) Composite outcome measures of PK variables | over 32hours after administration
  Composite outcome measures of PK variables
Lung exposure of B17MP, Formoterol and Glycopyrronium bromide without charcoal block (To evaluate the lung exposure (as AUCt and Cmax) Composite outcome measures of PK variables | over 32hours after administration
  Composite outcome measures of PK variables

SECONDARY OUTCOMES:
Systemic effects of CHF5993 (To evaluate the systemic effects as potassium and glucose levels) Composite outcome measures of PD variables | over 24hours after administration
  Composite outcome measures of PD variables
Systemic cardiac effects and the general safety (Composite outcome measures of cardiac variables (such as HR, BP, QT) and safety variables (such as AE, SAE) | over 24hours after administration
  Composite outcome measures of cardiac variables (such as HR, BP, QT) and safety variables (such as AE, SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS CPU Antwerpen, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No